CLINICAL TRIAL: NCT03587311
Title: A Randomized Phase 2 Study of Bevacizumab and Either Weekly Anetumab Ravtansine or Weekly Paclitaxel in Platinum-Resistant or Platinum Refractory Ovarian Cancer
Brief Title: Bevacizumab and Anetumab Ravtansine or Paclitaxel in Treating Patients With Refractory Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-01503; NCI-2018-01503 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHL-098; 10150 (Other: University Health Network Princess Margaret Cancer Center LAO); 10150 (Other: CTEP); UM1CA186644 (NIH)
Record Dates: First submitted 2018-07-13; First posted 2018-07-16 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube High Grade Serous Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian High Grade Serous Adenocarcinoma; Platinum-Resistant Fallopian Tube Carcinoma; Platinum-Resistant Ovarian Carcinoma; Platinum-Resistant Primary Peritoneal Carcinoma; Primary Peritoneal High Grade Serous Adenocarcinoma
MeSH Terms: interventions — anetumab ravtansine; Bevacizumab; Immunoglobulin G; Disulfides; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GROUP I (anetumab ravtansine, bevacizumab) (Experimental): Patients receive anetumab ravtansine IV over 1 hour on days 1, 8, 15, and 22 and bevacizumab over 30-90 minutes IV on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anetumab Ravtansine; Biological: Bevacizumab
- GROUP II (paclitaxel, bevacizumab) (Experimental): Patients receive paclitaxel on days 1, 8, 15, and 22 and bevacizumab over 30-90 minutes IV on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Paclitaxel

INTERVENTIONS:
Biological: Anetumab Ravtansine — Given IV
  Other Names: BAY 94-9343
  Arms: GROUP I (anetumab ravtansine, bevacizumab)
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: GROUP II (paclitaxel, bevacizumab)

SUMMARY:
This phase II trial studies the side effects of bevacizumab and anetumab ravtansine or paclitaxel in treating patients with ovarian, fallopian tube, or primary peritoneal cancer that does not respond to treatment (refractory). Bevacizumab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. Anetumab ravtansine is a drug that targets a protein in the body called mesothelin, which can be found in some ovarian, pancreatic and other tumors. Chemotherapy drugs, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether giving bevacizumab and anetumab ravtansine or paclitaxel may work better in treating patients with ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of the combination of weekly anetumab ravtansine (anetumab) and bi-weekly bevacizumab.

II. To determine whether the progression free survival (PFS) of the combination weekly anetumab and bi-weekly bevacizumab is superior to weekly paclitaxel and bi-weekly bevacizumab.

SECONDARY OBJECTIVES:

I. To determine the overall response rate (ORR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1.

II. To evaluate the pharmacokinetic (PK) profiles of weekly anetumab in serum and in peripheral blood mononuclear cells (PBMCs).

III. To evaluate anti-drug antibody (ADA) titers (only for patients receiving anetumab).

IV. To evaluate mononuclear phagocyte system (MPS) function, Fc-gamma receptors (FcgammaRs), hormone and chemokine mediators.

V. To correlate the expression of CA125 (immunohistochemistry [IHC] & serum) with mesothelin expression in archival tissue and circulating megakaryocyte potentiating factor (MPF).

VI. To investigate blood-based angiome profiling as a potential biomarker. VII. To characterize the molecular profile of archival tumor tissue using the Oncomine panel, and explore whether genomic mutations such as BRCA1/2 and homologous repair deficiency status are associated with clinical outcome.

EXPLORATORY OBJECTIVE:

I. To assess tumor tissue-based VEGF-dependent gene expression signature as a biomarker of response.

OUTLINE:

PHASE I: Patients receive anetumab ravtansine intravenously (IV) over 1 hour on days 1, 8, 15, and 22 and bevacizumab over 30-90 minutes IV on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive anetumab ravtansine and bevacizumab as in Phase I.

GROUP II: Patients receive paclitaxel on days 1, 8, 15, and 22 and bevacizumab over 30-90 minutes IV on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30-37 days and then every 8 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed high grade serous or high grade endometrioid ovarian, fallopian tube, primary peritoneal cancer
* Patients must have platinum resistant (platinum-free interval < 6 months) or platinum refractory disease as per Gynecological Cancer Intergroup (GCIC) criteria
* Patients must have radiologic evidence of disease progression
* Criteria only for the randomized phase 2 part: patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3 x 10^9/L
* Absolute neutrophil count >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Total bilirubin =< upper limit of normal (ULN) (except in Gilbert's syndrome)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (ULN)
* Serum creatinine =< 1.5 x ULN OR creatinine clearance >= 50 mL/min/1.73 m^2 for patients with creatinine levels above 1.5 x institutional normal (using the Cockcroft Gault formula)
* Urine protein / creatinine ratio (UPCR) =< 1
* Ongoing prior toxicities related to previous treatments must be recovered to < grade 2 at the time of registration (with the exception of alopecia, grade 2 peripheral neuropathy or lymphopenia)
* Criteria only for the randomized phase 2 part: mesothelin screen positive determined from archival tumor tissue and to be performed centrally. MSLN-positive is defined as >= 30% of tumor cells with membrane staining intensities >= 2+. If an archival tumor specimen is unavailable, or unsuitable for mesothelin testing, a pre-treatment fresh tumor biopsy is required

  * For the run-in-phase 1, patients will not be selected based on the mesothelin expression
* Patients with known brain metastases are not excluded from this clinical trial. Patients who received palliative radiation (for brain metastases) are eligible if they have been asymptomatic for at least 4 weeks without use of maintenance steroid therapy, and last received radiation at least 4 weeks prior to proposed start of therapy
* Ability to understand and the willingness to sign a written informed consent document. Patients with Impaired Decision Making Capacity (IDMC) can have a Legally Authorized Representative sign on their behalf. Documentation, such as a Power of Attorney, must be presented in order for a substitute decision maker to be allowed

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients who are receiving any other investigational agents
* History of severe allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab, anetumab ravtansine or paclitaxel
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list or medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product. Strong inhibitors and inducers of CYP3A4 are prohibited within 2 weeks before the start of and during treatment. Strong inhibitors and inducers of CYP2C8 should be used with caution; the PI of the study is to be consulted regarding their use
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued during the study and for at least 6 months after last dose of study drugs. These potential risks may also apply to other agents used in this study. Women of child-bearing potential who do not agree to use adequate contraceptive measures during study therapy and for at least 6 months after the completion of study therapy will be excluded. Should a patient become pregnant or suspect she is pregnant while she is participating in this study, the patient should inform the treating physician immediately
* Serious or non-healing wound, ulcer or bone fracture
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to day 1
* Invasive procedures defined as follows:

  * Major surgical procedure or significant traumatic injury within 28 days prior to day 1 therapy, or open biopsy within 7 days prior to day 1 therapy
  * Anticipation of need for major surgical procedures during the course of the study
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to day 1
* Patients with clinically significant cardiovascular disease are excluded

  * Inadequately controlled hypertension (HTN) (systolic blood pressure [SBP] > 160 mmHg and/or diastolic blood pressure [DBP] > 90 mmHg despite antihypertensive medication)
  * History of cerebrovascular accident (CVA) within 6 months
  * Myocardial infarction or unstable angina within 6 months
  * Serious and inadequately controlled cardiac arrhythmia
  * Significant vascular disease (e.g. aortic aneurysm, history of aortic dissection)
  * Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Current symptom of keratitis or retinopathy at >= grade 2
* Resting electrocardiogram (ECG) with corrected QT interval by Fridericia (QTcF) > 470 msec or family history of long QT syndrome
* History of bowel obstruction within 28 days from proposed start of treatment
* History or evidence of arterial thrombotic or hemorrhagic disorders within 3 months before proposed start of treatment, non-healing wound, ulcer, or bone fracture
* Prior use of weekly paclitaxel or bevacizumab in the platinum resistant (disease progression within 6 months of platinum based chemotherapy)/refractory (disease progression during or following the 3 months of the first line platinum based chemotherapy) setting
* Known active human immunodeficiency virus (HIV) or hepatitis B or C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2018-10-12 (Actual); Primary Completion 2026-10-21 (Estimated); Study Completion 2026-10-21 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From the time of treatment start assessed up to 1 year
  PFS will be estimated using the Kaplan-Meier method and compared between groups with log rank test. Summary statistics will be provided, such as the median, 6-month and estimates, along with 95% confidence intervals. Plots will also be constructed which show the PFS estimate and 95% confidence intervals.

SECONDARY OUTCOMES:
Response rate assessed using Response Evaluation Criteria in Solid Tumors | Up to 1 year
  Only one, single, final analysis is planned and statistical significance will be defined at the alpha = 0.05 level. All tests will be two-sided and 95% confidence levels will be constructed for outcomes of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lheureux, Principal Investigator — University Health Network Princess Margaret Cancer Center LAO
Locations (23):
- United States (22):
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - HaysMed, Hays, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada